CLINICAL TRIAL: NCT03437772
Title: Third Generation Cognitive Behavioural Therapy Versus Treatment-as-usual for Attention Deficit and Hyperactivity Disorder: a Randomized, 2-parallel-group, Evaluator Blinded, Superiority Trial
Brief Title: Third Generation Cognitive Behavioural Therapy vs Treatment-as-usual for ADHD
Acronym: Hyper-mCBT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: PHRC-N/2016/JLC-01
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Adhd
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CBT with mindfulness
  Interventions: Behavioral: Mindfulness Cognitive Behavioral Therapy program
- Treatment as Usual: Barkley therapy

INTERVENTIONS:
Behavioral: Mindfulness Cognitive Behavioral Therapy program — 16 simultaneous-but-separate therapy sessions for parents and children.
  Groups: CBT with mindfulness

SUMMARY:
The investigators hypothesize that the mindfulness Cognitive Behavioral Therapy program will lead to a reduction in attention deficit and hyperactivity disorder symptoms, anxiety and depression, and improve self-confidence, emotional control, social integration and school results.

ELIGIBILITY:
Inclusion Criteria:

* If deemed able, the patient must have given his/her informed and signed consent
* The parents (or legal guardian) of minor patients must have given their informed and signed consent.
* The patient and participating parents must be insured or beneficiary of a health insurance plan
* The patient is equal to or greater than 7 years old and less than or equal to 15 years old
* The patient presents with attention deficit and hyperactivity disorder with an ADHDRS-PI score > 27
* The patient is currently not under treatment - OR - is treated with methylphenidate with a stable posology (not expected to vary in the near future) but remains symptomatic

Exclusion Criteria:

* The patient is participating in, or has participated in over the past three months, another trial or another study that may interfere with the results or conclusion of the present study
* The patient is in an exclusion period determined by a previous study
* The participating parent(s) is(are) under judicial protection, or is an adult under guardianship
* It is impossible to correctly inform the patient or his/her parent or legal guardian
* Patients or parents refusing participation, signature of the signed consent or follow-up procedures
* Previously documented mental retardation (IQ < 70) or suspicion thereof by the investigator
* The patient has already participated in cognitive behavioural therapy (individual or group) in the six months preceding inclusion
* Patients diagnosed with autism spectrum disorder, psychotic disorder or bipolar disorder
* The family has participated in a parental guidance programme in the last 6 months.
* The family has already participated in the present study

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Families consulting for attention deficit and hyperactivity disorder
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
ADHD symptom severity | baseline
  clinical-rated ADHD rating scale (ADHDRS-PI) questionnaire; score ranges 0-54
ADHD symptom severity | Month 5
  clinical-rated ADHD rating scale (ADHDRS-PI) questionnaire; score ranges 0-54
ADHD symptom severity | Month 8
  clinical-rated ADHD rating scale (ADHDRS-PI) questionnaire; score ranges 0-54

SECONDARY OUTCOMES:
Parenting styles | Baseline
  Parental Authority Questionnaire (PAQ); 30 items per parent
Parenting styles | Month 5
  Parental Authority Questionnaire (PAQ); 30 items per parent
Parenting styles | Month 8
  Parental Authority Questionnaire (PAQ); 30 items per parent
The quality of life for parents. | Baseline
  Parental - Developmental Disorders - Quality of Life (PAR-DD-QoL) questionnaire; score ranges from 17-85
The quality of life for parents. | Month 5
  Parental - Developmental Disorders - Quality of Life (PAR-DD-QoL) questionnaire; score ranges from 17-85
The quality of life for parents. | Month 8
  Parental - Developmental Disorders - Quality of Life (PAR-DD-QoL) questionnaire; score ranges from 17-85
Global function | Baseline
  Clinical Global Impression Scale (CGI-S) questionnaire; score from 1-7
Global function | Month 5
  Clinical Global Impression Scale (CGI-S) questionnaire; score from 1-7
Global function | Month 8
  Clinical Global Impression Scale (CGI-S) questionnaire; score from 1-7
Global function | Baseline
  Children's Global Assessment Scale CGAS) questionnaire; score ranges from 0-100
Global function | Month 5
  Children's Global Assessment Scale CGAS) questionnaire; score ranges from 0-100
Global function | Month 8
  Children's Global Assessment Scale CGAS) questionnaire; score ranges from 0-100
Social well-being and school parameters for children | Baseline
  CONNERS for school teachers; cut-off for significant behavioral problem >15 his questionnaire will be given to the first patients included to 149 th patient included
Social well-being and school parameters for children | Baseline
  SDQ ; cut-off for significant behavioral problem >15 . his questionnaire will be given to the first patients included to 149 th patient included his questionnaire will be given to 150th patients included to 248th patient included
Social well-being and school parameters for children | Month 5
  SDQ ; cut-off for significant behavioral problem >15 . his questionnaire will be given to the first patients included to 149 th patient included his questionnaire will be given to 150th patients included to 248th patient included
Social well-being and school parameters for children | Month 8
  CONNERS for school teachers; cut-off for significant behavioral problem >15 his questionnaire will be given to the first patients included to 149 th patient included
Anxiety in children | Baseline
  Multidimensional Anxiety Scale for Children (MASC) questionnaire; 39-item, 4-point Likert scale
Anxiety in children | Month 5
  Multidimensional Anxiety Scale for Children (MASC) questionnaire; 39-item, 4-point Likert scale
Anxiety in children | Month 8
  Multidimensional Anxiety Scale for Children (MASC) questionnaire; 39-item, 4-point Likert scale
Depression in children | Baseline
  Children depression inventory (CDI) questionnaire; score ranges from 0-54
Depression in children | Month 5
  Children depression inventory (CDI) questionnaire; score ranges from 0-54
Depression in children | Month 8
  Children depression inventory (CDI) questionnaire; score ranges from 0-54
Anxiety and depression in parents | Baseline
  Hospital Anxiety and Depression Scale (HADS) questionnaire; 2 subscores each ranging from 0-21
Anxiety and depression in parents | Month 5
  Hospital Anxiety and Depression Scale (HADS) questionnaire; 2 subscores each ranging from 0-21
Anxiety and depression in parents | Month 8
  Hospital Anxiety and Depression Scale (HADS) questionnaire; 2 subscores each ranging from 0-21
Self-Esteem and behaviour for children. | Baseline
  Rosenberg scale; score ranges from 0-40
Self-Esteem and behaviour for children. | Month 5
  Rosenberg scale; score ranges from 0-40
Self-Esteem and behaviour for children. | Month 8
  Rosenberg scale; score ranges from 0-40
Self-Esteem and behaviour for children. | Baseline
  CONNERS questionnaire for parents; cut-off for significant behavioral problem >15
Self-Esteem and behaviour for children. | Month 5
  CONNERS questionnaire for parents; cut-off for significant behavioral problem >15
Self-Esteem and behaviour for children. | Month 8
  CONNERS questionnaire for parents; cut-off for significant behavioral problem >15

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Lopez Castroman, M.D, Principal Investigator — CHU Nimes
Locations (4):
- France (4):
  - CHU Montpellier, Montpellier
  - CHU Nimes, Nîmes
  - APHP - Hôpital Robert Debré, Paris
  - Chu de Strasbourg, Strasbourg

REFERENCES:
- [Derived] Crouzet L, Gramond A, Suehs C, Fabbro-Peray P, Abbar M, Lopez-Castroman J. Third-generation cognitive behavioral therapy versus treatment-as-usual for attention deficit and hyperactivity disorder: a multicenter randomized controlled trial. Trials. 2022 Jan 28;23(1):83. doi: 10.1186/s13063-021-05983-2. PMID 35090544